CLINICAL TRIAL: NCT00002509
Title: HIGH-DOSE CHEMOTHERAPY WITH CYCLOPHOSPHAMIDE, ETOPOSIDE, AND CARBOPLATIN FOLLOWED BY RESCUE WITH AUTOLOGOUS BONE MARROW AND AUTOLOGOUS PERIPHERAL BLOOD STEM CELLS IN PATIENTS WITH POOR PROGNOSIS BREAST CANCER
Brief Title: High-Dose Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Poor-Prognosis Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Temple University Bone Marrow Transplant Program, Temple University Health Systems
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078064; TUHSC-1992; NCI-V92-0205
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Etoposide; Mesna; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: mesna
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining peripheral stem cell transplantation with combinations of drugs may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of high-dose combination chemotherapy followed by peripheral stem cell transplantation or autologous bone marrow transplantation in women with stage II breast cancer with eight or more positive axillary lymph nodes and in women with stage III or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Investigate the curative potential of high-dose cyclophosphamide, etoposide, and carboplatin followed by autologous stem cell rescue in women with breast cancer considered incurable by conventional therapy. II. Observe the overall response rate, survival rate, and toxicity associated with this regimen.

OUTLINE: Prior to therapy, patients undergo collection of peripheral blood stem cells (PBSC) on another protocol; patients with marrow involvement undergo PBSC harvest only, while all others may also undergo bone marrow harvest. All patients receive cyclophosphamide, etoposide, and carboplatin over 4 consecutive days, followed 3 days later by PBSC or bone marrow and granulocyte colony-stimulating factor. Patients are followed for duration of remission and survival.

PROJECTED ACCRUAL: 100-200 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed invasive (stage II-IV) carcinoma of the breast 8 or more positive axillary nodes required for stage II disease Chemotherapy-responsive disease required of patients with measurable or evaluable disease Partial or complete response to 3 courses of standard cyclophosphamide/doxorubicin/fluorouracil (CAF) or, for patients who have had CAF, cyclophosphamide/methotrexate/fluorouracil (CMF) 3-month course of standard mitomycin/vinblastine or paclitaxel acceptable in patients clearly resistant to CAF or CMF Visceral response despite progression in bone will be considered on an individual basis Patients with no evidence of disease may be entered without evidence of a chemotherapy response Resectable disease must be surgically removed prior to transplantation Hormone receptor status: If estrogen-receptor positive, prior failure with at least 1 hormonal manipulation required unless patient is premenopausal or has rapidly progressing visceral disease No more than 20% of marrow involved with tumor

PATIENT CHARACTERISTICS: Age: 15 to 60 Sex: Women only Menopausal status: Not specified Performance status: Karnofsky 80%-100% Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL AST less than 2 times normal Albumin at least 3.0 g/dL Renal: Creatinine less than 1.8 mg/dL BUN less than 20 mg/dL Cardiovascular: Left ventricular ejection fraction at least 55% Pulmonary: DLCO, FEV1, and FVC at least 50% of predicted pO2 at least 70 mm Hg on room air Other: No serious psychiatric, neurologic, or medical illness that would compromise the safety of a bone marrow transplant Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: See Disease Characteristics Radiotherapy: No prior chest irradiation other than to locally involved lymph nodes Surgery: See Disease Characteristics

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1991-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Klumpp, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Temple University Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Klumpp TR, Goldberg SL, Mangan KF, et al.: High dose cyclophosphamide, etoposide, and carboplatin (CEC) with autologous stem cell rescue for chemosensitive metastatic and high risk breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 13: A-245, 111, 1994.